CLINICAL TRIAL: NCT06145152
Title: Using AI-generated Adaptive Training Recommendations to Improve Physical Performance
Brief Title: Adaptive Training Recommendations for Improved Physical Performance
Acronym: ELLIDA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Swedish School of Sport and Health Sciences (Other)
Collaborators: Silicon Valley Exercise Analytics (svexa) (Unknown)
Responsible Party: Principal Investigator, Filip Larsen, Associate Professor, The Swedish School of Sport and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Ellida
Record Dates: First submitted 2023-11-06; First posted 2023-11-22 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Maximal Oxygen Consumption; Physical Performance
Keywords: exercise; AI
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive (Experimental): Subjects in the Adaptive group will get updated and adjusted training programs based on daily readiness level
  Interventions: Procedure: Adaptive exercise training
- Static (Active Comparator): Subjects in the Static group will get the same inital training program as the Adaptive group but will not get updated and adjusted training programs based on daily readiness level
  Interventions: Procedure: Static exercise training

INTERVENTIONS:
Procedure: Adaptive exercise training — The training recommendation for the day will be adjusted based on the readiness level. The adjustments can be both up or down (increased or decreased training)
  Arms: Adaptive
Procedure: Static exercise training — The training recommendation for the day will not be adjusted based on the readiness level.
  Arms: Static

SUMMARY:
In this study two different training strategies are compared; one is adaptive where the training is adjusted up or down on a daily basis to better match the recovery status (readiness) of the subject. The other strategy is static, i.e. no changes are made depending on readiness level. Instead the subjects in the static group are encouraged to perform the prescribed training.

The training intervention will last for 8 weeks.

Thorough physiological tests will be performed pre and post the training intervention together with muscle biopsies for assessment of mitochondrial function.

DETAILED DESCRIPTION:
40 recreational athletes, 20 male and 20 females, will be recruited to this study. The research subjects will be stratified into two groups: an Adaptive and a Static training group. The training sessions will be mainly home-based training according to daily instructions from an online application. Testing sessions will be performed on a laboratory treadmill. During the entire period (run-in + training period) the participants will wear continuous glucose monitors for minute-by-minute glucose tracking, an Oura ring for sleep measurements, a Garmin GPS watch with heart rate chest-strap for training data and answer questiions regarding subjective well-being using an online application (Readiness Advisor).

The training program will be a mixture of training sessions based on the experience levels of the research subject.

During the onboarding session, data from each persons Garmin watch, will be used to create an optimal training program that takes into account recent training history and which type of training each subject responds the best to. For the subjects in the Adaptive group the training will be adjusted up or down on a daily basis based on subjective readiness, sleep or glucose control. The subjects in the Static group will not get any adjustments in their training program regardless of readiness level.

The length of the training intervention will be 8 weeks.

In addition to adjusting the training for the adaptive group based on daily readiness, the training in that group will be adjusted based on actual training done. For example if a participant fails to reach his suggested heart rate range during a prescribed session, the training load for upcoming sessions will be recalculated so that the weekly overall training load goal is achieved. This kind of adjustments will not be done in the static training group.

Both pre and post the training period a battery of physiological tests will be done including determination of VO2max, lactate threshold and running economy. A performance test (3000m time-trial) will be done on a running track.

A muscle biopsy will be donated from the Vastus Lateralis for assessment of mitochondrial function, efficiency, capacity and density using a combination of methods including respirometry, western blot and enzymatic methods. Capillarization and number of myonuclei will be assessed using histochemical staining. In addition muscle buffering capacity will be investigated using an acid-titration assay.

In addition to the physiological and biochemical investigation, parameters such as subjective training tolerability, perceived pleasure of the training and number of dropouts are important objectives in the proposed studie.

Statistical power calculation. Based on the parallel group design, 80% power, an alpha of 0.05 and a coefficient of variation of 2.4% for VO2max, 4.2% for performance and 14% for mitochondrial function, a differences can be detected between groups of 6%, 11% and 26% for the three outcomes if 15 participants per group are included. 20 subjects will be recruited per group to allow for 5 dropouts per group.

ELIGIBILITY:
Inclusion Criteria:

* Training history of at least two running sessions per week (5km +) the last 6 months
* No chronic diseases
* Able to perform maximal exercise
* Having used a smart watch for training frequently during the last 3 months
* Willing to use wearable technology (Oura ring, continuous glucose monitor, running GPS watch)

Exclusion Criteria:

* Heart, lung or metabolic disease
* Recurrent running injuries
* Not willing to use wearable devices
* Performing a subtantial amount of non-running exercise training

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Physical performance | pre intervention and within 5 days post intervention
  3000 meter time trial performance

SECONDARY OUTCOMES:
Maximal oxygen consumption | pre intervention and within 5 days post intervention
  maximal oxygen consumption at the end of an incremental exercise stress test
Lactate threshold | pre intervention and within 5 days post intervention
  lactate threshold (anaerobic threshold) as assessed by blood lactate concentration during a submaximal running test on the treadmill

CONTACTS AND LOCATIONS:
Locations (1):
- Swedish School of Sports and Health Sciences, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No